CLINICAL TRIAL: NCT02972697
Title: Evaluation of 11C-acetate PET Imaging as a Novel Approach to Detecting Pathology in Pulmonary TB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11C_acetate
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2016-11

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 11C-acetate PET (Experimental): 11C-acetate and FDG PET/MRI and PET/CT will be performed.
  Interventions: Radiation: 11C-acetate ligand; Radiation: FDG ligand

INTERVENTIONS:
Radiation: 11C-acetate ligand
Radiation: FDG ligand

SUMMARY:
Imaging using 11C-acetate PET (positron emission tomography) in patients with tuberculosis (TB) may be able to detect non-replicating persister bacilli. This may permit identification of those patients at risk of relapse following completion of TB treatment. The main aim of this pilot study is to assess the ability of 11C-acetate PET to detect pulmonary lesions in individuals with active pulmonary TB.

DETAILED DESCRIPTION:
Novel biomarkers for detecting pulmonary TB and response to treatment are sorely needed. PET in conjunction with either CT (computed tomography) or MRI (magnetic resonance imaging) scanning allows assessment of the metabolic activity of lesions as well as the structural anatomy of the lung. The standard radiolabelled tracer for PET is 18F-fluorodeoxyglucose (FDG) which labels metabolically active cells. However, one of the main limitations of FDG is the non-specific uptake leading to difficulty differentiating between tumours, infection and inflammatory pathologies.

11C-acetate is a PET ligand used currently to image various conditions but has not been used to identify TB lesions previously. 11C-acetate may be taken up by the lipid bodies in the dormant bacteria in TB, enabling visualization of this sub-population of bacteria. Using the 11C-acetate ligand for imaging pulmonary TB may add to the utility of PET scanning, potentially allowing monitoring of drug activity against the persister population and identification of those patients who may be at risk of relapse following drug therapy.

This pilot study will compare 11C-acetate to the standard ligand, FDG, using PET/CT and PET/MRI. The target population for this study is those individuals with confirmed pulmonary TB who have a high chance of demonstrable bacillary burden who are therefore likely to have populations of persister bacteria in the lungs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years and above
2. Willing to comply with the study visits and procedures
3. Willing and able to provide written informed consent
4. Clinical diagnosis of pulmonary TB with characteristic symptoms and compatible X-ray findings plus microbiological confirmation with one or more of (i) Acid-fast bacilli (AFB) smear-positive or (ii) molecular test positive or (iii) TB culture positive. Tests done at any time during the current episode of TB are acceptable for diagnostic purposes
5. Not on TB treatment or have completed less than 8 weeks of TB treatment

Exclusion Criteria:

1. Diabetes that is, in the judgment of the investigator, so poorly controlled that it would prevent adequate PET scanning
2. Cardiac pacemaker, aneurysm clip or other metallic implant considered unsafe for MRI
3. Known chronic kidney disease
4. Occupation involving substantial exposure to radiation
5. History of medical procedures in the last year involving substantial exposure to radiation (>2mSv)
6. Malignancy requiring chemotherapy or radiation
7. Women who are currently pregnant or breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value (SUV) of 11C-acetate PET in pulmonary TB lesions | Within 8 weeks of starting TB treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore